CLINICAL TRIAL: NCT05235269
Title: A Multicenter, Open-label, Single-arm, Phase 2 Study to Evaluate Safety and Organ Uptake Quantitation Repeatability of 124I AT-01 Using Positron Emission Tomography/X-ray Computed Tomography (PET/CT) in Subjects With Systemic Amyloidosis
Brief Title: A Study to Evaluate Organ Level Uptake Repeatability of 124I AT-01 in Subjects With Systemic Amyloidosis
Acronym: AT01-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Attralus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AT01--001
Record Dates: First submitted 2021-12-10; First posted 2022-02-11 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis
Keywords: Amyloid light chain (AL); Amyloid Transthyretin Systemic Amyloidosis (ATTR)
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Intervention Model Description: Single arm, no placebo, no comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): 124I-AT-01
  Interventions: Drug: 124I-AT-01

INTERVENTIONS:
Drug: 124I-AT-01 — All participants received 1 mCi 124I-AT-01 on Day 1 and at Week 6 via IV infusion over 2-5 minutes or slow IV bolus at 1 mL/5 seconds.
  Other Names: AT-01; I124-AT-01

SUMMARY:
This study is designed to assess the repeatability of organ-specific quantitation of radiotracer uptake following Positron Emission Tomography/Computed Tomography (PET/CT) imaging of AT- 01 in subjects with amyloid light chain (AL) or amyloid transthyretin (ATTR) systemic amyloidosis.

DETAILED DESCRIPTION:
This is a multicenter, open label, single arm study in subjects with amyloid light chain (AL) or amyloid transthyretin (ATTR) systemic amyloidosis with visceral amyloid deposits. This study consists of a screening period of up to 30 days; two one-day treatment periods (Day 1 and Week 6); a safety follow-up 24-48 hours after the second administration of 124I AT-01, and a safety follow-up visit 28 days after the second administration of 124I-AT-01.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the study procedures and is capable of giving signed informed consent, as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male or female ≥18 years of age.
3. For women of childbearing potential: agreement to remain abstinent or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 90 days after the last dose of 124I-AT-01.

   1. A woman is considered of childbearing potential if she is postmenarchal, has not reached a postmenopausal state, and has not undergone surgical sterilization.
   2. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
   3. Contraception methods that do not result in a failure rate of <1% per year such as cap, diaphragm, or sponge with spermicide, or male or female condom with or without spermicide, are not acceptable.
   4. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
4. For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

   a) With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 120 days (a spermatogenesis cycle) after the last dose of study intervention. Men must refrain from donating sperm during this same time period.
5. Able to undergo two PET/CT scans as part of the study, including ability to lie supine for up to 1 hour.
6. Has a history of AL or ATTR systemic amyloidosis with at least one organ with clinically demonstrable amyloid involvement defined by:

   1. AL systemic amyloidosis: Positive tissue biopsy for AL amyloid, and achieved a hematologic very good partial response or complete response based on their most recent assessment, and at least one of the following: 1) Organ biopsy positive for amyloid, or 2) Natriuretic peptide (NT-proBNP) >650 pg/mL, or 3) left ventricle septal wall thickness >12 mm by echocardiogram or cardiac magnetic resonance (CMR), or 4) 24-hour urine protein >500 mg, or 5) Urine albumin-to-creatinine ratio >300 mg/g
   2. ATTR (wild type or variant) systemic amyloidosis: Positive cardiac biopsy for ATTR amyloid, or at least two of the following: 1) Positive extracardiac tissue biopsy for ATTR amyloid or positive transthyretin gene mutation associated with amyloid, or 2) left ventricle septal wall thickness >12 mm by echocardiogram or CMR, or 3) pyrophosphate (PYP) scintigraphy with myocardial uptake ≥grade 2.

Exclusion Criteria

1. Is pregnant or breast-feeding.
2. Is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of psychosis.
3. Has received in the last 6 months or are currently receiving treatment with anti-amyloid monoclonal antibody therapy or are expected to begin treatment prior to completing this study.
4. Has received heparin or heparin analogs within 7 days of Day 1.
5. Has a significant co-morbidity (e.g., Easter Cooperative Oncology Group (ECOG) score of 3 or greater), New York Heart Association (NYHA) Class IV heart failure, uncontrolled infection, or other ongoing serious illness.
6. Has active thyroid disease.
7. Has a known allergy to potassium iodine treatment.
8. Is receiving hemodialysis or peritoneal dialysis.
9. Has severe claustrophobia that would prevent completion of the PET/CT imaging protocol.
10. Has received an investigational agent within five half-lives of the agent or 30 days, whichever is longer, prior to Screening.
11. Has any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M. Bell, MD, Study Director — Attralus, Inc.
Locations (3):
- United States (3):
  - PET/CT Imaging of Berkeley, Berkeley, California
  - Northern California PET Imaging Center, Sacramento, California
  - PET/CT Imaging of San Jose, San Jose, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the initial 34 participants screened, 32 participants met inclusion criteria and were enrolled for treatment. Two participants were screen failures, one of whom was re-screened and subsequently enrolled in the study.
Period: Overall Study
Arm/Group | 124I-AT-01
Started | 33
Day 1 | 33
Week 6 | 27
Safety Follow-up 1 | 26
Safety Follow-up 2 (EOS) | 26
Completed | 26
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Participant elected to drop out (i.e., not undergo second scan) but did not withdraw consent | 1
Not completed — Protocol-specified withdrawal criterion met | 5

BASELINE CHARACTERISTICS:
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Within-Participant Coefficient of Variation [wCV] Associated With the Quantification (SUVmax) of Radioactivity Associated With Organ-Level Radiotracer Uptake
Description: Between-visit repeatability of organ-specific (heart, kidney, liver, spleen) quantitation (SUVmax) of radiotracer uptake following PET/CT imaging of 124I-AT-01 in participants with AL or ATTR systemic amyloidosis was assessed.
  wCV with its associated 95% RC provides guidance on the level of change in organ-specific quantitation of radiotracer uptake that needs to be observed to be confident that a true change in uptake has occurred. Smaller values of wCV represent better agreement. Computation of wCV and associated RCs in addition to the two-sided 95% CI is described in the SAP.
  Only images from participants/organs with positive uptake were included. RCs between visits were calculated using the difference of the log of the average of the 2 reads for a reader at Day 1 and the log of the average of the 2 reads for the same reader at Week 6. The 95% RCs were calculated on the log-transformed data and exponentiated to determine the limits in percentages.
Time Frame: Day 1 and Week 6
Population: The Image Evaluable Set was defined as all participants who underwent PET/CT scans on both Day 1 and 6 to 8 weeks after Day 1 and who had evaluable images at both time points.
Measure: Number (95% Confidence Interval); unit: coefficient of variation
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 27
coefficient of variation
  Heart - Reader 1: number analyzed (Participants) | 20
  Heart - Reader 1 | 14.58 [-31.4 to 45.8]
  Heart - Reader 2: number analyzed (Participants) | 20
  Heart - Reader 2 | 14.50 [-31.3 to 45.5]
  Heart - Reader 3: number analyzed (Participants) | 20
  Heart - Reader 3 | 12.97 [-28.7 to 40.2]
  Kidney - Reader 1: number analyzed (Participants) | 16
  Kidney - Reader 1 | 16.28 [-34.2 to 51.9]
  Kidney - Reader 2: number analyzed (Participants) | 16
  Kidney - Reader 2 | 9.46 [-22.2 to 28.5]
  Kidney - Reader 3: number analyzed (Participants) | 16
  Kidney - Reader 3 | 15.18 [-32.4 to 48.0]
  Liver - Reader 1: number analyzed (Participants) | 5
  Liver - Reader 1 | 14.38 [-31.1 to 45.1]
  Liver - Reader 2: number analyzed (Participants) | 5
  Liver - Reader 2 | 6.54 [-16.1 to 19.2]
  Liver - Reader 3: number analyzed (Participants) | 5
  Liver - Reader 3 | 7.97 [-19.1 to 23.7]
  Spleen - Reader 1: number analyzed (Participants) | 7
  Spleen - Reader 1 | 8.69 [-20.6 to 26.0]
  Spleen - Reader 2: number analyzed (Participants) | 7
  Spleen - Reader 2 | 9.64 [-22.5 to 29.1]
  Spleen - Reader 3: number analyzed (Participants) | 7
  Spleen - Reader 3 | 8.39 [-20.1 to 25.0]

2. Primary Outcome: Within-Participant Coefficient of Variation [wCV] Associated With the Quantification (SUVpeak) of Radioactivity Associated With Organ-Level Radiotracer Uptake
Description: Between-visit repeatability of organ-specific (heart, kidney, liver, spleen) quantification (SUVpeak) of radiotracer uptake following PET/CT imaging of 124I-AT-01 in participants with AL or ATTR systemic amyloidosis was assessed.
  wCV with its associated 95% RC provides guidance on the level of change in organ-specific quantitation of radiotracer uptake that needs to be observed to be confident that a true change in uptake has occurred. Computation of wCV and associated RCs in addition to the two-sided 95% CI is described in the SAP.
  Only images from participants/organs with positive uptake were included. RCs between visits were calculated using the difference of the log of the average of the 2 reads for a reader at Day 1 and the log of the average of the 2 reads for the same reader at Week 6. The 95% RCs were calculated on the log-transformed data and exponentiated to determine the limits in percentages.
Time Frame: Day 1 and Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: coefficient of variation
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 27
coefficient of variation
  Heart - Reader 1: number analyzed (Participants) | 20
  Heart - Reader 1 | 13.06 [-28.8 to 40.5]
  Heart - Reader 2: number analyzed (Participants) | 20
  Heart - Reader 2 | 11.57 [-26.2 to 35.5]
  Heart - Reader 3: number analyzed (Participants) | 20
  Heart - Reader 3 | 8.21 [-19.6 to 24.5]
  Kidney - Reader 1: number analyzed (Participants) | 16
  Kidney - Reader 1 | 12.82 [-28.4 to 39.7]
  Kidney - Reader 2: number analyzed (Participants) | 16
  Kidney - Reader 2 | 9.95 [-23.1 to 30.1]
  Kidney - Reader 3: number analyzed (Participants) | 16
  Kidney - Reader 3 | 13.88 [-30.2 to 43.4]
  Liver - Reader 1: number analyzed (Participants) | 5
  Liver - Reader 1 | 9.68 [-22.6 to 29.2]
  Liver - Reader 2: number analyzed (Participants) | 5
  Liver - Reader 2 | 8.37 [-20.0 to 25.0]
  Liver - Reader 3: number analyzed (Participants) | 5
  Liver - Reader 3 | 8.32 [-19.9 to 24.8]
  Spleen - Reader 1: number analyzed (Participants) | 7
  Spleen - Reader 1 | 12.47 [-27.8 to 38.5]
  Spleen - Reader 2: number analyzed (Participants) | 7
  Spleen - Reader 2 | 12.48 [-27.8 to 38.5]
  Spleen - Reader 3: number analyzed (Participants) | 7
  Spleen - Reader 3 | 12.84 [-28.4 to 39.8]

3. Primary Outcome: Intraclass Correlation Coefficient (ICC) Associated With the Quantification (SUVmax) of Radioactivity Associated With Organ-Level Radiotracer Uptake
Description: Repeatability of organ-specific (heart, kidney, liver, spleen) quantification (SUVmax) of radiotracer uptake following PET/CT imaging of 124I-AT-01 in participants with AL or ATTR systemic amyloidosis was assessed.
  ICC assesses the consistency or reproducibility of measurements made by the 3 readers measuring the same participant images.
  Reader results are the average of the reader's 2 reads for the specific visit. A two-way mixed effects model with absolute agreement type for a single rater/measurement was used to calculate the ICC. The ICC coefficient is the ratio of the between-cluster variance to the total variance (denoted as r in the SAP). Fisher's z-transformation was used to calculate the 95% confidence intervals. A two-sided 95% CI is computed based upon the formulary provided in the SAP.
Time Frame: Day 1 and Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 27
correlation coefficient
  Heart - Day 1 | 0.903 [0.796 to 0.955]
  Heart - Week 6 | 0.955 [0.903 to 0.980]
  Kidney - Day 1 | 0.973 [0.940 to 0.988]
  Kidney - Week 6 | 0.964 [0.922 to 0.984]
  Liver - Day 1 | 0.971 [0.937 to 0.987]
  Liver - Week 6 | 0.975 [0.946 to 0.989]
  Spleen - Day 1 | 0.991 [0.979 to 0.996]
  Spleen - Week 6 | 0.996 [0.992 to 0.998]

4. Primary Outcome: Intraclass Correlation Coefficient (ICC) Associated With the Quantification (SUVpeak) of Radioactivity Associated With Organ-Level Radiotracer Uptake
Description: Repeatability of organ-specific (heart, kidney, liver, spleen) quantification (SUVpeak) of radiotracer uptake following PET/CT imaging of 124I-AT-01 in participants with AL or ATTR systemic amyloidosis was assessed.
  ICC assesses the consistency or reproducibility of measurements made by the 3 readers measuring the same participant images.
  Reader results are the average of the reader's 2 reads for the specific visit. A two-way mixed effects model with absolute agreement type for a single rater/measurement was used to calculate the ICC. The ICC coefficient is the ratio of the between-cluster variance to the total variance (denoted as r in the SAP). Fisher's z-transformation was used to calculate the 95% confidence intervals. A two-sided 95% CI is computed based upon the formulary provided in the SAP.
Time Frame: Day 1 and Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 27
correlation coefficient
  Heart - Day 1 | 0.960 [0.913 to 0.982]
  Heart - Week 6 | 0.987 [0.970 to 0.994]
  Kidney - Day 1 | 0.994 [0.986 to 0.997]
  Kidney - Week 6 | 0.991 [0.980 to 0.996]
  Liver - Day 1 | 0.993 [0.984 to 0.997]
  Liver - Week 6 | 0.990 [0.978 to 0.995]
  Spleen - Day 1 | 0.997 [0.992 to 0.998]
  Spleen - Week 6 | 0.999 [0.997 to 0.999]

5. Secondary Outcome: Number of Participants With At Least 1 Treatment-Emergent Adverse Event (TEAE)
Description: TEAEs were defined as events that were newly reported or reported to worsen in severity after the start of treatment. Adverse events (AEs) that occurred after the treatment start date, occurred on the treatment start date with a time that was equal to or after treatment start time, or that had a missing AE start date were categorized as treatment emergent.
Time Frame: Day 1 through the end of the study (up to 14 weeks)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Count of Participants; unit: Participants
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
Participants | 13

6. Secondary Outcome: Clinical Laboratory Values - Chemistry (mmol/L)
Description: Changes from baseline in chemistry clinical laboratory values with units of mmol/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
mmol/L
  Calcium - Week 6: number analyzed (Participants) | 27
  Calcium - Week 6 | -0.028 (0.1079)
  Calcium - Safety Follow-up 1: number analyzed (Participants) | 25
  Calcium - Safety Follow-up 1 | -0.035 (1.1013)
  Carbon Dioxide - Week 6: number analyzed (Participants) | 27
  Carbon Dioxide - Week 6 | -0.7 (3.06)
  Carbon Dioxide - Safety Follow-up 1: number analyzed (Participants) | 25
  Carbon Dioxide - Safety Follow-up 1 | -1.0 (2.29)
  Chloride - Week 6: number analyzed (Participants) | 27
  Chloride - Week 6 | -0.9 (2.65)
  Chloride - Safety Follow-up 1: number analyzed (Participants) | 25
  Chloride - Safety Follow-up 1 | 0.4 (2.74)
  Glucose - Week 6: number analyzed (Participants) | 27
  Glucose - Week 6 | 0.3515 (1.34157)
  Glucose - Safety Follow-up 1: number analyzed (Participants) | 25
  Glucose - Safety Follow-up 1 | 0.1310 (1.63653)
  Phosphate - Week 6: number analyzed (Participants) | 26
  Phosphate - Week 6 | 0.0025 (0.16570)
  Phosphate - Safety Follow-up 1: number analyzed (Participants) | 24
  Phosphate - Safety Follow-up 1 | 0.0229 (0.16665)
  Potassium - Week 6: number analyzed (Participants) | 27
  Potassium - Week 6 | -0.11 (0.462)
  Potassium - Safety Follow-up 1: number analyzed (Participants) | 25
  Potassium - Safety Follow-up 1 | 0.4 (2.74)
  Sodium - Week 6: number analyzed (Participants) | 27
  Sodium - Week 6 | -0.2 (3.32)
  Sodium - Safety Follow-up 1: number analyzed (Participants) | 25
  Sodium - Safety Follow-up 1 | 0.8 (2.71)
  Urea Nitrogen - Week 6: number analyzed (Participants) | 27
  Urea Nitrogen - Week 6 | 0.2116 (1.81616)
  Urea Nitrogen - Safety Follow-up 1: number analyzed (Participants) | 25
  Urea Nitrogen - Safety Follow-up 1 | -0.0429 (2.17049)

7. Secondary Outcome: Clinical Laboratory Values - Chemistry (Umol/L)
Description: Changes from baseline in chemistry clinical laboratory values with units of umol/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
umol/L
  Bilirubin - Week 6: number analyzed (Participants) | 27
  Bilirubin - Week 6 | 1.0136 (4.00446)
  Bilirubin - Safety Follow-up 1: number analyzed (Participants) | 25
  Bilirubin - Safety Follow-up 1 | 1.2315 (2.44487)
  Creatinine - Week 6: number analyzed (Participants) | 27
  Creatinine - Week 6 | 5.24 (18.541)
  Creatinine - Safety Follow-up 1: number analyzed (Participants) | 25
  Creatinine - Safety Follow-up 1 | 1.77 (14.430)

8. Secondary Outcome: Clinical Laboratory Values - Chemistry (g/L)
Description: Changes from baseline in chemistry clinical laboratory values with units of g/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
g/L
  Albumin - Week 6: number analyzed (Participants) | 27
  Albumin - Week 6 | -0.4 (2.79)
  Albumin - Safety Follow-up 1: number analyzed (Participants) | 25
  Albumin - Safety Follow-up 1 | -1.5 (2.84)
  Protein - Week 6: number analyzed (Participants) | 27
  Protein - Week 6 | -0.7 (4.22)
  Protein - Safety Follow-up 1: number analyzed (Participants) | 25
  Protein - Safety Follow-up 1 | -1.7 (3.61)

9. Secondary Outcome: Clinical Laboratory Values - Chemistry (IU/L)
Description: Changes from baseline in chemistry clinical laboratory values with units of IU/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
IU/L
  Alanine Aminotransferase - Week 6: number analyzed (Participants) | 27
  Alanine Aminotransferase - Week 6 | -1.4 (9.54)
  Alanine Aminotransferase - Safety Follow-up 1: number analyzed (Participants) | 25
  Alanine Aminotransferase - Safety Follow-up 1 | -2.6 (8.03)
  Alkaline Phosphatase - Week 6: number analyzed (Participants) | 27
  Alkaline Phosphatase - Week 6 | -2.9 (13.20)
  Alkaline Phosphatase - Safety Follow-up 1: number analyzed (Participants) | 25
  Alkaline Phosphatase - Safety Follow-up 1 | -3.1 (12.46)
  Aspartate Aminotransferase - Week 6: number analyzed (Participants) | 27
  Aspartate Aminotransferase - Week 6 | -0.3 (6.78)
  Aspartate Aminotransferase - Safety Follow-up 1: number analyzed (Participants) | 25
  Aspartate Aminotransferase - Safety Follow-up 1 | -1.8 (5.64)
  Lactate Dehydrogenase - Week 6: number analyzed (Participants) | 27
  Lactate Dehydrogenase - Week 6 | 1.1 (55.16)
  Lactate Dehydrogenase - Safety Follow-up 1: number analyzed (Participants) | 25
  Lactate Dehydrogenase - Safety Follow-up 1 | -6.0 (49.70)

10. Secondary Outcome: Clinical Laboratory Values - Hematology (% of White Blood Cell [WBC] Count)
Description: Changes from baseline in hematology clinical laboratory values with units of % of WBC count
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: % of WBC count
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
% of WBC count
  Basophils/Leukocytes - Week 6: number analyzed (Participants) | 26
  Basophils/Leukocytes - Week 6 | -0.1 (0.77)
  Basophils/Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Basophils/Leukocytes - Safety Follow-up 1 | -0.1 (0.81)
  Eosinophils/Leukocytes - Week 6: number analyzed (Participants) | 26
  Eosinophils/Leukocytes - Week 6 | -0.2 (1.41)
  Eosinophils/Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Eosinophils/Leukocytes - Safety Follow-up 1 | -0.1 (1.72)
  Lymphocytes/Leukocytes - Week 6: number analyzed (Participants) | 26
  Lymphocytes/Leukocytes - Week 6 | 0.0 (6.62)
  Lymphocytes/Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Lymphocytes/Leukocytes - Safety Follow-up 1 | 1.1 (6.32)
  Monocytes/Leukocytes - Week 6: number analyzed (Participants) | 26
  Monocytes/Leukocytes - Week 6 | -0.3 (4.57)
  Monocytes/Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Monocytes/Leukocytes - Safety Follow-up 1 | -0.7 (4.68)
  Neutrophils/Leukocytes - Week 6: number analyzed (Participants) | 26
  Neutrophils/Leukocytes - Week 6 | 0.6 (9.62)
  Neutrophils/Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Neutrophils/Leukocytes - Safety Follow-up 1 | -0.1 (9.59)

11. Secondary Outcome: Clinical Laboratory Values - Hematology (10^9 Cells/L)
Description: Changes from baseline in hematology clinical laboratory values with units of 10^9 cells/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
10^9 cells/L
  Basophils - Week 6: number analyzed (Participants) | 26
  Basophils - Week 6 | -0.02 (0.051)
  Basophils - Safety Follow-up 1: number analyzed (Participants) | 22
  Basophils - Safety Follow-up 1 | -0.03 (0.057)
  Eosinophils - Week 6: number analyzed (Participants) | 26
  Eosinophils - Week 6 | -0.02 (0.085)
  Eosinophils - Safety Follow-up 1: number analyzed (Participants) | 22
  Eosinophils - Safety Follow-up 1 | -0.01 (0.108)
  Leukocytes - Week 6: number analyzed (Participants) | 26
  Leukocytes - Week 6 | -0.27 (1.961)
  Leukocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Leukocytes - Safety Follow-up 1 | -0.29 (2.115)
  Lymphocytes - Week 6: number analyzed (Participants) | 26
  Lymphocytes - Week 6 | -0.02 (0.314)
  Lymphocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Lymphocytes - Safety Follow-up 1 | 0.02 (0.287)
  Monocytes - Week 6: number analyzed (Participants) | 26
  Monocytes - Week 6 | -0.02 (0.208)
  Monocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Monocytes - Safety Follow-up 1 | -0.06 (0.156)
  Neutrophils - Week 6: number analyzed (Participants) | 26
  Neutrophils - Week 6 | -0.22 (1.984)
  Neutrophils - Safety Follow-up 1: number analyzed (Participants) | 22
  Neutrophils - Safety Follow-up 1 | -0.21 (2.028)
  Platelets - Week 6: number analyzed (Participants) | 26
  Platelets - Week 6 | 4.4 (35.43)
  Platelets - Safety Follow-up 1: number analyzed (Participants) | 22
  Platelets - Safety Follow-up 1 | 3.1 (37.26)

12. Secondary Outcome: Clinical Laboratory Values - Hematology (10^12 Cells/L)
Description: Changes from baseline in hematology clinical laboratory values with units of 10^12 cells/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
10^12 cells/L
  Erythrocytes - Week 6: number analyzed (Participants) | 26
  Erythrocytes - Week 6 | 0.000 (0.2684)
  Erythrocytes - Safety Follow-up 1: number analyzed (Participants) | 22
  Erythrocytes - Safety Follow-up 1 | -0.055 (0.2600)

13. Secondary Outcome: Clinical Laboratory Values - Hematology (g/L)
Description: Change from baseline in hematology clinical laboratory values with units of g/L
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
g/L
  Hemoglobin - Week 6: number analyzed (Participants) | 26
  Hemoglobin - Week 6 | -0.4 (8.60)
  Hemoglobin - Safety Follow-up 1: number analyzed (Participants) | 22
  Hemoglobin - Safety Follow-up 1 | -2.1 (8.28)

14. Secondary Outcome: Clinical Laboratory Values - Hematology (% of Total Blood Cell Count)
Description: Changes from Baseline in hematology clinical laboratory values with units of % of total blood cell count
Time Frame: At Week 6 and Safety Follow-up 1 (24 to 48 hours after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: % of total blood cell count
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
% of total blood cell count
  Hematocrit - Week 6: number analyzed (Participants) | 26
  Hematocrit - Week 6 | -0.19 (2.554)
  Hematocrit - Safety Follow-up 1: number analyzed (Participants) | 22
  Hematocrit - Safety Follow-up 1 | -0.54 (2.521)

15. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure (mmHg)
Description: Changes from baseline in blood pressure measurements with units of mmHg
Time Frame: Day 1 post-administration and Week 6 pre-administration and post-administration
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
mmHg
  Systolic Blood Pressure - Day 1 Post-Administration: number analyzed (Participants) | 20
  Systolic Blood Pressure - Day 1 Post-Administration | -2.8 (9.21)
  Systolic Blood Pressure - Week 6 Pre-Administration: number analyzed (Participants) | 27
  Systolic Blood Pressure - Week 6 Pre-Administration | -3.9 (15.97)
  Systolic Blood Pressure - Week 6 Post-Administration: number analyzed (Participants) | 26
  Systolic Blood Pressure - Week 6 Post-Administration | -8.5 (16.98)
  Diastolic Blood Pressure - Day 1 Post-Administration: number analyzed (Participants) | 20
  Diastolic Blood Pressure - Day 1 Post-Administration | -3.2 (6.65)
  Diastolic Blood Pressure - Week 6 Pre-Administration: number analyzed (Participants) | 27
  Diastolic Blood Pressure - Week 6 Pre-Administration | 0.2 (11.01)
  Diastolic Blood Pressure - Week 6 Post-Administration: number analyzed (Participants) | 26
  Diastolic Blood Pressure - Week 6 Post-Administration | -2.2 (11.45)

16. Secondary Outcome: Change From Baseline in Vital Signs - Heart Rate (Beats/Min)
Description: Changes from baseline in heart rate measurements with units of beats/min
Time Frame: Day 1 post-administration and Week 6 pre-administration and post-administration
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
beats/min
  Heart Rate - Day 1 Post-Administration: number analyzed (Participants) | 20
  Heart Rate - Day 1 Post-Administration | 1.1 (7.93)
  Heart Rate - Week 6 Pre-Administration: number analyzed (Participants) | 27
  Heart Rate - Week 6 Pre-Administration | 0.9 (7.37)
  Heart Rate - Week 6 Post-Administration: number analyzed (Participants) | 26
  Heart Rate - Week 6 Post-Administration | 1.0 (7.21)

17. Secondary Outcome: Change From Baseline in Anti-Drug Antibodies (ADA)
Description: Changes from baseline in ADA
Time Frame: Post-dose at Week 6 or Safety Follow-up 2 (28 days after Week 6)
Population: The Safety Set was defined as all participants who received any amount of 124I-AT-01.
Measure: Count of Participants; unit: Participants
Arm/Group | 124I-AT-01
Number analyzed (Participants) | 33
Participants
  Negative for ADA at Screening and negative for ADA post-dose: number analyzed (Participants) | 26
  Negative for ADA at Screening and negative for ADA post-dose | 26
  Negative for ADA at Screening and positive for ADA post-dose: number analyzed (Participants) | 26
  Negative for ADA at Screening and positive for ADA post-dose | 0

ADVERSE EVENTS:
Time Frame: Time of informed consent until the end of the study (up to 14 weeks)
Arm/Group | 124I-AT-01
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 124I-AT-01 (N=33)
Thalamic infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 124I-AT-01 (N=33)
Chest discomfort (General disorders) | 2
Oedema peripheral (General disorders) | 1
Vessel puncture site bruised (General disorders) | 1
COVID-19 (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dysponea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Blood lactic acid increase (Investigations) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data will be regarded as confidential until analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented at scientific meetings by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor. Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee, for comment.

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT05235269/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT05235269/SAP_001.pdf